CLINICAL TRIAL: NCT06192420
Title: Multi-centre, Double-blind, Randomised, Active- and Placebo-Controlled, Confirmatory Trial to Demonstrate Efficacy and Safety of Traumed® Gel in Patients Having Acute Ankle Sprain
Brief Title: TRAUMED - a Clinical Trial in Acute Ankle Sprain
Acronym: TRAUMED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biologische Heilmittel Heel GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C1502; 2016-004792-50 (EudraCT Number)
Record Dates: First submitted 2021-08-17; First posted 2024-01-05 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2021-08

CONDITIONS: Ankle Sprain
Keywords: Double blind clinical trial; Active and placebo controlled clinical trial; Leg injury
MeSH Terms: conditions — Ankle Injuries; Motor Activity; Leg Injuries | interventions — Traumeel S

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, active- and placebo-controlled confirmatory clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: CRO (including CRAs)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test product (Experimental): Traumed® gel (human gel galenic form of Traumeel®)
  Interventions: Drug: Traumeel®
- Reference product (Active Comparator): Diclofenac sodium gel 1%
  Interventions: Drug: Diclofenac sodium gel 1%
- Placebo therapy (Placebo Comparator): Corresponding placebo gel
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Traumeel® — 3g of gel three times daily for 7days (+1 day visit window)
  Other Names: Traumed® gel
  Arms: Test product
Drug: Diclofenac sodium gel 1% — 3g of gel three times daily for 7days (+1 day visit window)
  Other Names: Diclofenac Heumann gel
  Arms: Reference product
Drug: Placebo — 3g of gel three times daily for 7days (+1 day visit window)
  Other Names: Placebo gel
  Arms: Placebo therapy

SUMMARY:
TRAUMED - a randomized clinical trial evaluating the efficacy and safety of Traumed® gel in patients with acute ankle sprain.

DETAILED DESCRIPTION:
Lateral ankle sprains are the most prevalent musculoskeletal injuries in physically active populations. They also have a high prevalence in the general population and pose a substantial healthcare burden. The injury mechanism is characterized by a high velocity inversion and internal rotation of the ankle/foot complex. The treatment for acute lateral ankle sprain is quite variable, with many patients returning to activity in a short period of time; however, half of the affected population may never seek initial care. Inadequate treatment of ankle sprains can lead to chronic problems such as decreased range of motion, pain, and joint instability.

Controlled trials of Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) in patients with ankle sprain showed that compared with placebo, NSAIDs were associated with improved pain control and function, decreased swelling, and more rapid return to activity. Diclofenac is meanwhile considered to be the gold standard in the treatment of joint sprains and other conditions. Topical diclofenac is well tolerated and is associated with fewer side-effects than other topical NSAIDs, mostly mild, easily resolved local skin irritation.

The current trial is designed to demonstrate the superior efficacy of Traumed® gel versus placebo and to assess the non-inferiority of Traumed® gel compared to diclofenac gel. After evaluation of entry criteria patients will be randomized to investigational treatment, which will be Traumed® gel or diclofenac gel or matching placebo gel, administered locally on the area of the injury, 3 times daily for 7 days. After end of the 7-day treatment phase patients will be followed up for another 7 days. Consequently the entire duration of the trial for each patient will be 14 days.

Patients will receive paracetamol (acetaminophen) 500 mg/tablets as rescue medication to be taken for pain relief when necessary.

All patients will receive soft support (elastic bandage). Grade 2 patients will receive a semi-rigid removable brace on Day 7.

Primary and secondary outcomes are listed separately as required. All statistical tests will be two-sided with a significance level of alpha =0.05, unless specified otherwise.

Confirmatory analyses

1. Area Under the Curve (AUC) for pain on passive movement in Visual Analog Scale (VAS) from Baseline to Day 4 (test for superiority, Traumed® gel versus placebo), Full Analysis Set (FAS).
2. AUC for pain on passive movement in VAS from Baseline to Day 4 (test for non-inferiority, Traumed® gel versus diclofenac gel), Per-Protocol (PP) analysis set.

If the first a priori ordered test (superiority) shows statistical significance, the subsequent hypothesis (non-inferiority) can then be tested individually in a confirmatory manner according to the principle of a priori ordered hypotheses.

Clinical safety will be addressed by assessing Adverse Events (AEs), physical examinations, vital signs and as needed laboratory assessments in a descriptive manner.

Estimation of sample size is based on the primary efficacy variable, AUC for pain on passive movement as measured by VAS from Baseline to Day 4. A two-sided test of equality of the investigational drug (Traumed® gel) and the comparator (placebo) at level 0.05 based on an expected raw scale treatment difference of AUC 25 [mm x days] and a common standard deviation of AUC 75 [mm x days] for the response variables (re-expressed for nonparametric evaluation in terms of the Mann-Whitney (MW) statistic as MW = 0.6, achieves a power of at least 90% for parametric first line analysis as well as for second line nonparametric analysis if the sample size is set to 291 patients for the Traumed® gel group and to 146 patients for the placebo group.

Due to an additional safety requirement that AEs with incidence level of 1% for Traumed® gel are found during the trial with probability 95%, 299 patients for the Traumed® gel group are required. Assuming a drop-out rate from the Safety Analysis Set of about 4% an amount of 312 randomized patients in the Traumed® gel group is needed. With an allocation ratio of 2:1:1 (Traumed® gel : diclofenac gel : placebo gel) 156 patients are obtained in the diclofenac gel and placebo group each, that is, a total of 624 patients with acute unilateral Grade 1 or Grade 2 sprain of the lateral ankle.

During the recruitment phase site inspections by the German Local Authorities in 2019 (Gesundheitsamt Düsseldorf of German Federal State North Rhine Westphalia, NRW) it was recognized that there could have been a possible violation of the predefined 'blinding firewall' described in the protocol at some locations.

All sites were checked rigorously to detect any risk of unintentional deblinding, which, in the end, was not found. To exclude any risk of including these patients, the German regulatory authority (Federal Institute for Drugs and Medical Devices) recommended including only those cases in the final analysis where blinding could be 100% confirmed.

In order to ensure the pre-defined power of the trial for the trial objectives including the confirmatory test for non-inferiority (Traumed® gel compared to diclofenac gel), which is based on the Per-Protocol Analysis Set (PP), a sample size enhancement is introduced for compensation of cases for whom maintenance of blinding procedures may have been compromised and, thus, are representing a major protocol violation (exclusion from PP analysis).

For compensation, the final sample size will be enhanced to 202 patients for the diclofenac and Placebo group each, and to 404 patients for the Traumed® gel group resulting in a new total of 808 patients .

Analyses will be based on the Safety Analysis, Full Analysis, and the Per-Protocol analysis sets. The definitions of the analysis sets follow those given in the ICH E9 guideline (CMP/ICH/363/96).

ELIGIBILITY:
Inclusion Criteria:

* Acute unilateral Grade 1 or Grade 2 sprain of the lateral ankle.
* >/=18 years of age.
* Legally competent male or female outpatient.
* Injury occurred within previous 24 hours before first treatment expected.
* Signed Informed Consent.
* After 5 minutes of rest, pain on passive movement by investigator measured by Visual Analog Scale (VAS) >50 mm.
* Not pregnant or breast-feeding.

Exclusion Criteria:

* Similar injury affecting the same joint within the past 6 months.
* Bilateral ankle injury.
* Grade 3 ankle sprain.
* Fracture of the ankle (It should be excluded by using e.g., the Ottawa Ankle Rules. In case of any doubt the exclusion of fracture by x-ray should be considered as per standard of care).
* Chronic joint disorders such as clinically relevant osteoarthritis or aseptic arthritis
* Disorders that may lead to joint oedema for other reasons than ankle sprain (such as heart failure, thrombosis, lymphedema and others).
* Diagnosis requiring bed rest, hospitalization, surgery, or use of any cast during the planned treatment period.
* Debilitating acute or chronic illness.
* Use of systemic and /or topical corticosteroids in the previous 8 weeks, any analgesics (e.g., paracetamol / acetaminophen) in the previous 24 hours before Screening Visit, or 48 hours in the case of long-acting NSAID, cyclooxygenase type 2 (COX-2) specific inhibitors, or tramadol and other opioids. Low dose acetylsalicylic acid (70 - 100 mg per day) for anti-thrombotic therapy is permitted if doses are stable for the month prior to Screening Visit and planned to be stable during the entire study.
* History of sensitivity to any component of the study drugs (including e.g. paracetamol / acetaminophen intolerance; patients in whom asthma attacks, skin rash or acute rhinitis are triggered by acetylsalicylic acid or non-steroidal anti-inflammatory drugs (NSAIDs).
* Unwilling or unable to comply with all the requirements of the study protocol.
* Concurrent injury to proximal structures in ipsilateral lower extremity (i.e., concurrent shin, knee, thigh, or hip injury).
* History of ligament avulsion, fracture or surgery to the affected lower extremity.
* Presence of infections and/or skin diseases in the area of the study treatment site (including psoriasis).
* Any previous treatments of the injured ankle, whether topical or systemic, are prohibited except RICE (simultaneous combination of all 4 elements; Rest, Ice, Compression and Elevation; which is restricted to be used until starting treatment with the investigational drug).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 809 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC)* for pain on passive movement in Visual Analog Scale (VAS) from Baseline to Day 4. | Baseline and Day 4
  Ankle pain is assessed via a 100 mm VAS, where zero mm indicates 'no pain' and 100 mm indicates the 'most severe imaginable pain' in relation to the participant's ankle sprain. After 5 minutes rest, participants first assess their ankle sprain pain on a 100 mm VAS for a secondary efficacy assessment. With the participant still at rest, the investigator performs 10° dorsal-flexion and 30° plantar-flexion of the sprained ankle, before participants re-assess their pain on a 100 mm VAS.
Area Under the Curve (AUC) for pain on passive movement in Visual Analog Scale (VAS) from Baseline to Day 7 as per SAP version 1.0. | Baseline and Day 7
  Ankle pain is assessed via a 100 mm VAS, where zero mm indicates 'no pain' and 100 mm indicates the 'most severe imaginable pain' in relation to the participant's ankle sprain. After 5 minutes rest, participants first assess their ankle sprain pain on a 100 mm VAS for a secondary efficacy assessment. With the participant still at rest, the investigator performs 10° dorsal-flexion and 30° plantar-flexion of the sprained ankle, before participants re-assess their pain on a 100 mm VAS.

SECONDARY OUTCOMES:
AUC for pain at rest in VAS from Baseline to Day 4. | Baseline and Day 4
  Ankle pain is assessed via a 100 mm VAS, where zero mm indicates 'no pain' and 100 mm indicates the 'most severe imaginable pain' in relation to the participant's ankle sprain. After 5 minutes rest, participants assess their ankle sprain pain on a 100 mm VAS.
AUC for pain on passive movement in VAS from Baseline to Day 2, 7 and Final Visit. | Baseline, Day 2, Day 7 and Day 14
  Ankle pain is assessed via a 100 mm VAS, where zero mm indicates 'no pain' and 100 mm indicates the 'most severe imaginable pain' in relation to the participant's ankle sprain. After 5 minutes rest, participants assess their ankle sprain pain on a 100 mm VAS. With the participant still at rest, the investigator performs 10° dorsal-flexion and 30° plantar-flexion of the sprained ankle, before participants re-assess their pain on a 100 mm VAS.
AUC for pain at rest in VAS from Baseline to Day 2, 7 and Final Visit. | Baseline, Day 2, Day 7 and Day 14
  Ankle pain is assessed via a 100 mm VAS, where zero mm indicates 'no pain' and 100 mm indicates the 'most severe imaginable pain' in relation to the participant's ankle sprain. After 5 minutes rest, participants assess their ankle sprain pain on a 100 mm VAS.
Change from Baseline of pain on passive movement in VAS to Day 4, 7 and Final Visit. | Baseline, Day 4, Day 7 and Day 14
  Ankle pain is assessed via a 100 mm VAS, where zero mm indicates 'no pain' and 100 mm indicates the 'most severe imaginable pain' in relation to the participant's ankle sprain. After 5 minutes rest, participants assess their ankle sprain pain on a 100 mm VAS. With the participant still at rest, the investigator performs 10° dorsal-flexion and 30° plantar-flexion of the sprained ankle, before participants re-assess their pain on a 100 mm VAS.
Change from Baseline of pain at rest in VAS to Day 4, 7 and Final Visit. | Baseline, Day 4, Day 7 and Day 14
  Ankle pain is assessed via a 100 mm VAS, where zero mm indicated 'no pain' and 100 mm indicates the 'most severe imaginable pain' in relation to the participant's ankle sprain. After 5 minutes rest, participants assess their ankle sprain pain on a 100 mm VAS.
Change from Baseline to Day 2, 4, 7 and Final Visit in the Foot and Ankle Ability Measure (FAAM) Activities of Daily Living (ADL) sub-scale. | Baseline, Day 2, Day 4, Day 7 and Day 14
  The FAAM questionnaire allows self-reported assessment of physical function of participants with musculoskeletal disorders of the leg, foot, and ankle. The FAAM-ADL sub-scale, which is part of the FAAM questionnaire, consists of 21 items assessing Activities of Daily Living (ADL) including standing, walking, going up stairs, etc. Participants in this trial assess difficulty in performing ADL by answering; 'no difficulty', 'slight difficulty', 'moderate difficulty', 'extreme difficulty', 'unable to do' or 'not applicable'. The response to each item on the FAAM-ADL sub-scale is recorded from 4 'no difficulty' to 0 'unable to do'. For each participant, the total score will be multiplied by 100/84 (84 = highest potential score) such that final scores are standardized to a 0 to 100 score, where 0 = worst physical function and 100 = best physical function.
Amount of rescue medication (doses) required for pain relief. | Baseline, Day 4, Day 7 and Day 14
  Participant use of rescue medication is reported in participant diaries and rescue medication drug accountability forms throughout the trial. Paracetamol (acetaminophen), 500 mg/tablet is permitted when necessary for pain with a maximum of 4 tablets or 2,000 mg/day (but not more than 2 tablets at a time). Participants are not allowed to take paracetamol within 8 hrs prior to Day 2 visit or within 24 hrs of visits at days 4, 7 and 14. The number of Paracetamol tablets taken by a participant up to each participant visit will be reported.
Time to 50% improvement of pain at rest measured by VAS at participant visits. | Baseline through to Day 14
  The time to 50% improvement will be calculated from the VAS assessments of pain at rest performed at all participant visits using the percent changes from Baseline (recorded at Day 1).
To assess the tolerability and safety of Traumed® gel as measured by the number of participants experiencing Adverse Events. | From signature of Informed consent (Day 1) to Final Visit (Day 14)
  All Adverse Events (AEs) that occur during the entire course of the trial after the participant has signed the informed consent will be collected and reported, regardless of whether they are reported by the participant, elicited by investigator questioning, detected through physical examination, or by other means. These will include AEs observed at the site of administration of the investigational drug (lateral ankle). AE intensity is determined by the investigator as Mild, Moderate or Severe, based on his/her direct observations or the participant's reporting for AEs occurring in between participant visits.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Becker, Prof,PhD,MD, Principal Investigator — UKSH Universitätsklinikum Schleswig-Holstein, Campus Kiel
Locations (1):
- UKSH Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerdesmeyer L, Pabst H, Cesnulevicius K, Schultz M, Smit A, Kerkhoffs G. Tr14 gel for the treatment of acute ankle sprains: a plain language summary of the TRAUMED trial. J Comp Eff Res. 2025 Jul;14(7):e250018. doi: 10.57264/cer-2025-0018. Epub 2025 Jun 5. PMID 40468690

DOCUMENTS (2):
  • Study Protocol (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT06192420/Prot_002.pdf
  • Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/20/NCT06192420/SAP_003.pdf